CLINICAL TRIAL: NCT06083844
Title: Phase II Investigation of Pembrolizumab in Combination With Bevacizumab and Oral Cyclophosphamide in Patients With High Grade Ovarian Cancer and Surgically Documented Minimal Residual Disease After Frontline Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0685; NCI-2023-08686 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pembrolizumab; Bevacizumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab in Combination with Bevacizumab and Oral Cyclophosphamide (Experimental): Participants will begin receiving the study drug Pembrolizumab in Combination with Bevacizumab and Oral Cyclophosphamide.
  Each study cycle is 21 days.
  Interventions: Drug: Pembrolizumab; Drug: Bevacizumab; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Pembrolizumab — Given by IV (vein)
  Other Names: KEYTRUDA®
Drug: Bevacizumab — Given by IV (vein)
  Other Names: Avastin™; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Cyclophosphamide — Given by mouth
  Other Names: Cytoxan®; Neosar®

SUMMARY:
To find out if combining pembrolizumab, bevacizumab (or an equivalent biosimilar drug), and low-dose cyclophosphamide can help control high-grade ovarian cancer that has MRD after treatment. The safety of this treatment combination will also be studied.

DETAILED DESCRIPTION:
Primary Objectives

1. To determine whether the combination of pembrolizumab, bevacizumab (or equivalent biosimilars) and oral low dose cyclophosphamide can improve PFS by 6 months (compared to historical control/current trial) in patients with high grade ovarian cancer with residual disease identified by second look laparoscopy.

Secondary Objectives

1. To determine the safety of the above regimen in this patient population.

Exploratory Objectives

1. Correlating clinical benefit with gene expression and immune profiles of tumor tissue from SLL and confirmatory biopsy at the time of radiological progression.
2. Tumor cell free tumor DNA (ctDNA) is emerging as a potentially sensitive marker of response in patients undergoing immunotherapy treatment(Lee et al. 2018). We will compare serial plasma ctDNA levels with response by RECIST v1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of high grade non-mucinous epithelial ovarian cancer will be enrolled in this study.
2. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 2 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 2 during the treatment period and for at least 120 days after the last dose of study medication.
3. The participant provides written informed consent for the trial.
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
5. Have received standard of care frontline surgical and chemotherapy treatment (at least six cycles of platinum and taxane (or equivalent, with or without bevacizumab/biosimilar therapy). Patients who received neoadjuvant therapy are included. Omission of one or more doses of chemo for toxicity or hypersensitivity reaction is allowed. Have minimal residual disease (MRD) after a complete clinical response to frontline therapy (defined as: having a normalization of CA-125 and no obvious evidence of disease on exam or imaging unless the patient has an elevated CA-125 thought to be due to other confounding causes by the treating physician). Imaging with subtle or indeterminate findings will not disqualify participation.
6. Having MRD is defined as either of the following conditions (must occur within 3 months on the last dose of frontline platinum-taxane chemotherapy):

   1. Second-look surgery that may be performed either as standard of care or in the context of a non-therapeutic clinical trial with positive tissue or cytology.

      OR
   2. Detectable ctDNA by the Signatera assay. Assay results that are "positive below analytical range" qualify as detectable.
7. Participants who have undergone second look surgery, must have histologically confirmed residual ovarian cancer at time of second-look surgery. Patients with cytological evidence of malignant cells in washings obtained as part of the second look procedure are eligible even if biopsies are negative.
8. Be willing to allow use of archival tissue from second-look surgery (if performed) and primary surgery or biopsy for use in this study.
9. Have adequate organ function as determined by the following laboratory values:

   1. ANC ≥ 1,000 /mcL
   2. Platelets ≥ 100,000 / mcL
   3. Hgb ≥8 g/dL (transfusion allowed)
   4. Creatinine Clearance ≥30 mL/min (measured or calculated per local practice)
   5. Total Bilirubin ≤ 1.5 × ULN or ≤ 3 × ULN in the case of suspected/documented Gilbert's Syndrome
   6. AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN
10. Have adequately recovered from second look surgery to be able to start the investigational regimen no sooner than 28 days from the date of second look surgery, and within 7 weeks of this procedure.
11. Negative serum pregnancy test within 72 hours prior to receiving the first dose of study medication (unless surgically sterile or postmenopausal for greater than one year).

Exclusion Criteria:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
2. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
3. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
4. Is currently receiving or has received an investigational agent within 4 weeks prior to the first dose of study intervention.
5. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. Steroids to reduce risk of radiologic contrast allergy is permitted.
6. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
7. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, type I diabetes mellitus, etc.) is not considered a form of systemic treatment and is allowed.
9. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
10. Serious active infection that in the opinion of treating physician would preclude participation.
11. Has a known history of uncontrolled Human Immunodeficiency Virus (HIV) infection. Patients with normal CD4 count and undetectable viral load will be eligible.
12. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection that is active and has not been cured. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding or expecting to conceive children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
16. Has had an allogenic tissue/solid organ transplant.
17. Clinically significant uncontrolled hypertension as defined by SBP>150 or DBP>90 persistently documented within 30 days of starting study directed treatment. Patients would be eligible if blood pressure controliscontrol is achieved with appropriate anti-hypertensive therapy. Rescreening after this therapy has been instituted is allowed.
18. Histology showing mucinous or low-grade epithelial ovarian carcinoma.
19. Documented deleterious germline or somatic BRCA mutations or tumors known to be homologous recombination deficiency (HRD) positive (e.g. as determined by MyChoice by Myriad Genetics (or other CLIA certified labs per PI's discretion).
20. History of arterial thrombosis (pulmonary embolism in pulmonary arteries do not count as arterial thrombosis). Patients with history of DVT are eligible as long as they have received or are receiving appropriate anticoagulation therapy.
21. History of gastrointestinal or urinary fistulae, non-healed or chronic wound, or other conditions that, in the investigator's view, would contraindicate or significantly increase the risks of bevacizumab/biosimilar therapy.
22. Unable to understand or to comply with the study instructions and requirements or has a history of non-compliance to the medical regimen.
23. Concurrent or planned use of any other anti-cancer systemic chemotherapy, biological therapy (including hormonal or immune therapy), radiation therapy, or live cancer vaccines.

24 Any other medical condition that in the investigator's judgement would significantly increase the risks of the investigational regimen.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Jazaeri, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org